CLINICAL TRIAL: NCT00322972
Title: Eliminating Trachoma With Repeat Mass Drug Treatment
Brief Title: Trachoma Amelioration in Northern Amhara (TANA)
Acronym: TANA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Thomas M. Lietman, Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-02576
Record Dates: First submitted 2006-05-05; First posted 2006-05-09 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Trachoma; Chlamydia
Keywords: Bacterial Infections; Chlamydia Infections; Eye Diseases
MeSH Terms: conditions — Trachoma; Chlamydia Infections; Bacterial Infections; Eye Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- A (Other): Annual mass treatment
  Interventions: Drug: Mass treatment with oral azithromycin to an entire community
- B (Other): Biannual mass treatment
  Interventions: Drug: Mass treatment with oral azithromycin to an entire community
- C (Experimental): Mass administration of antibiotic; treatment of children (1-10 years of age) only
  Interventions: Drug: Mass treatment with oral azithromycin to an entire community
- D (No Intervention): Delayed initiation of mass administration of antibiotic
- F (Other): One-time mass administration only
  Interventions: Drug: Mass treatment with oral azithromycin to an entire community
- G (Experimental): One-time mass administration of antibiotics, plus intensive latrine construction
  Interventions: Drug: Mass treatment with oral azithromycin to an entire community

INTERVENTIONS:
Drug: Mass treatment with oral azithromycin to an entire community — For baseline and follow-up surveys prior to azithromycin distribution, a stratified random sample from two age groups will be chosen: 1) 60 study participants younger than 10 years old and 2) 60 study participants aged 10 years and above. Clinical examination will be performed and conjunctival swabs will be taken from all the study participants. For study arm C and D, nasopharyngeal swabs will be collected from 10 randomly selected children among the 60 participants under 10 who were recruited for conjunctival swabbing. Then a single dose of azithromycin will be distributed according to study design: in tablet form for adults; a weight-adjusted tablet dose for children ages 8-10; and pediatric suspension for children ages 1 - 7.
  Arms: A; B; C; F; G

SUMMARY:
The WHO has initiated a program to eliminate trachoma, blinding eye infection caused by Chlamydia trachomatis, in large part by mass distributions of oral azithromycin. The proposed study will determine the frequency and treatment target of community-wide mass antibiotic treatment. We will also study the impact of mass antibiotic distribution on antibiotic-resistance in pneumococcus.

DETAILED DESCRIPTION:
The proposed study is a group-randomized trial to determine the frequency and treatment target of community-wide mass antibiotic treatment to eliminate trachoma. We will also study the impact of community-wide antibiotic distribution on antibiotic-resistance in pneumococcus. Communities in Goncha Siso Enese district of East Gojam Zone, Ethiopia will be randomly assigned to different treatment schemes and monitored to study the following research questions:

Specific Aim 1. To determine whether biannual mass treatments is more likely to eliminate ocular chlamydia from hyper-endemic communities than annual mass treatments.

Specific Aim 2. To determine whether children form a core group for the transmission of trachoma.

Specific Aim 3. To determine whether latrine construction prevents the return of infection into a community after mass treatment.

Specific Aim 4. To determine the effect of mass azithromycin treatments on antibiotic resistance in pneumococcus and the reduction in mortality.

Specific Aim 5. To determine whether annual mass treatments are more likely to eliminate ocular chlamydia from hyper-endemic communities than biennial mass treatments.

ELIGIBILITY:
Inclusion Criteria:

• All residents residing in the state-teams which are randomly selected for this study.

Exclusion Criteria:

* Pregnant women
* Children under 6 months of age
* All those who are allergic to macrolides or azalides
* Refusal of village chief (for village inclusion), or refusal of parent or guardian (for individual inclusion)

Individuals in these three exclusion criteria will not be given the study antibiotic azithromycin, but offered the current WHO-recommended alternative treatment to azithromycin for active trachoma, which is 1% tetracycline eye ointment, to be used twice a day, topically to both eyes, for six weeks. Note that the exclusion criteria refer to the exclusion to the treatment drug, but not to the monitoring, treatment of trachoma, and examinations.

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 33000 (Actual)
Dates: Start 2006-06; Primary Completion 2009-11 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
The average prevalence of ocular chlamydia infection in communities in an arm as determined by pooled NAAT (Nucleic Acid Amplification Test)(at 42 months for Aim 1, at 12 months for Aim 2, post-treatment relative to pre-treatment for Aim 3) | 42 months

SECONDARY OUTCOMES:
Clinical active trachoma in community, as determined by the WHO simplified grading system | 42 months
Childhood (>= 1 year of age) mortality, analyzed as 1-5, 6-10 years of age, and total | 42 months
Macrolide resistance in pneumococcus (% resistance over time, clustered by randomization unit) | 42 months
Average prevalence of ocular chlamydia infection in annually and biennially treated communities as determined by pooled NAAT (Nucleic Acid Amplification Test) | 48 months
Diversity measure in the conjunctival and nasopharyngeal microbiomes of children (age 0-9) | 0, 6, 12, 18, 24, 30, 36, 42, and 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Tom Lietman, MD, Principal Investigator — Proctor Foundation, UCSF; Kieran S O'Brien, MPH, Study Director — Proctor Foundation, UCSF; Paul Emerson, PhD, Study Director — Emory University
Locations (1):
- Carter Center, Ethiopia, Addis Ababa, Ethiopia

REFERENCES:
- [Background] Skalet AH, Cevallos V, Ayele B, Gebre T, Zhou Z, Jorgensen JH, Zerihun M, Habte D, Assefa Y, Emerson PM, Gaynor BD, Porco TC, Lietman TM, Keenan JD. Antibiotic selection pressure and macrolide resistance in nasopharyngeal Streptococcus pneumoniae: a cluster-randomized clinical trial. PLoS Med. 2010 Dec 14;7(12):e1000377. doi: 10.1371/journal.pmed.1000377. PMID 21179434
- [Background] Porco TC, Gebre T, Ayele B, House J, Keenan J, Zhou Z, Hong KC, Stoller N, Ray KJ, Emerson P, Gaynor BD, Lietman TM. Effect of mass distribution of azithromycin for trachoma control on overall mortality in Ethiopian children: a randomized trial. JAMA. 2009 Sep 2;302(9):962-8. doi: 10.1001/jama.2009.1266. PMID 19724043
- [Background] Keenan JD, Ayele B, Gebre T, Zerihun M, Zhou Z, House JI, Gaynor BD, Porco TC, Emerson PM, Lietman TM. Childhood mortality in a cohort treated with mass azithromycin for trachoma. Clin Infect Dis. 2011 Apr 1;52(7):883-8. doi: 10.1093/cid/cir069. PMID 21427395
- [Background] Lietman TM, Gebre T, Ayele B, Ray KJ, Maher MC, See CW, Emerson PM, Porco TC; TANA Study Group. The epidemiological dynamics of infectious trachoma may facilitate elimination. Epidemics. 2011 Jun;3(2):119-24. doi: 10.1016/j.epidem.2011.03.004. Epub 2011 Apr 6. PMID 21624783
- [Background] Stoller NE, Gebre T, Ayele B, Zerihun M, Assefa Y, Habte D, Zhou Z, Porco TC, Keenan JD, House JI, Gaynor BD, Lietman TM, Emerson PM. Efficacy of latrine promotion on emergence of infection with ocular Chlamydia trachomatis after mass antibiotic treatment: a cluster-randomized trial. Int Health. 2011 Jun;3(2):75-84. doi: 10.1016/j.inhe.2011.03.004. PMID 21785663
- [Background] Keenan JD, See CW, Moncada J, Ayele B, Gebre T, Stoller NE, McCulloch CE, Porco TC, Gaynor BD, Emerson PM, Schachter J, Lietman TM. Diagnostic characteristics of tests for ocular Chlamydia after mass azithromycin distributions. Invest Ophthalmol Vis Sci. 2012 Jan 25;53(1):235-40. doi: 10.1167/iovs.11-8493. PMID 22159017
- [Background] Gebre T, Ayele B, Zerihun M, House JI, Stoller NE, Zhou Z, Ray KJ, Gaynor BD, Porco TC, Emerson PM, Lietman TM, Keenan JD. Latrine promotion for trachoma: assessment of mortality from a cluster-randomized trial in Ethiopia. Am J Trop Med Hyg. 2011 Sep;85(3):518-23. doi: 10.4269/ajtmh.2011.10-0720. PMID 21896815
- [Result] House JI, Ayele B, Porco TC, Zhou Z, Hong KC, Gebre T, Ray KJ, Keenan JD, Stoller NE, Whitcher JP, Gaynor BD, Emerson PM, Lietman TM. Assessment of herd protection against trachoma due to repeated mass antibiotic distributions: a cluster-randomised trial. Lancet. 2009 Mar 28;373(9669):1111-8. doi: 10.1016/S0140-6736(09)60323-8. PMID 19329003
- [Result] Gebre T, Ayele B, Zerihun M, Genet A, Stoller NE, Zhou Z, House JI, Yu SN, Ray KJ, Emerson PM, Keenan JD, Porco TC, Lietman TM, Gaynor BD. Comparison of annual versus twice-yearly mass azithromycin treatment for hyperendemic trachoma in Ethiopia: a cluster-randomised trial. Lancet. 2012 Jan 14;379(9811):143-51. doi: 10.1016/S0140-6736(11)61515-8. Epub 2011 Dec 20. PMID 22192488
- [Derived] Ray KJ, Zhou Z, Cevallos V, Chin S, Enanoria W, Lui F, Lietman TM, Porco TC. Estimating community prevalence of ocular Chlamydia trachomatis infection using pooled polymerase chain reaction testing. Ophthalmic Epidemiol. 2014 Apr;21(2):86-91. doi: 10.3109/09286586.2014.884600. PMID 24621121
- [Derived] Keenan JD, Ayele B, Gebre T, Moncada J, Stoller NE, Zhou Z, Porco TC, McCulloch CE, Gaynor BD, Emerson PM, Schachter J, Lietman TM. Ribosomal RNA evidence of ocular Chlamydia trachomatis infection following 3 annual mass azithromycin distributions in communities with highly prevalent trachoma. Clin Infect Dis. 2012 Jan 15;54(2):253-6. doi: 10.1093/cid/cir791. Epub 2011 Nov 17. PMID 22095569